CLINICAL TRIAL: NCT04592536
Title: A Randomized, Double-blind, Placebo- and Active Comparator-controlled, Crossover Trial to Examine the Effect of Multiple Doses of CVL-865 on Panic Symptoms Induced by Carbon Dioxide Inhalation in Healthy Subject
Brief Title: A Trial of the Effect of CVL-865 on Panic Symptoms Induced by Carbon Dioxide Inhalation in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cerevel Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVL-865-HV-001
Record Dates: First submitted 2020-09-29; First posted 2020-10-19 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Panic Disorder
Keywords: Anxiety; Panic; CVL-865; PF-06372865; Hypercapnia; CO2 challenge; Healthy Subjects
MeSH Terms: conditions — Panic Disorder; Anxiety Disorders; Hypercapnia | interventions — Alprazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CVL-865 (Experimental): High dose CVL-865 (25mg) Low dose CVL-865 (7.5mg)
  Interventions: Drug: CVL-865 High dose; Drug: CVL-865 low dose
- Alprazolam (Active Comparator): Active Comparator Alprazolam with extended release oral tablets; 1 tablet BID
  Interventions: Drug: Alprazolam 1mg XR
- Placebo (Placebo Comparator): Placebo Comparator matching oral tablets for CVL-865, capsule for Alprazolam
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CVL-865 High dose — High dose CVL-865: Will be administered as 5mg BID for 2 days followed by 12.5mg BID for another 2 days during the Titration Phase. 25mg will be administered during the Maintenance Phase (3 days of BID and morning dose only on the 4th day)
  Arms: CVL-865
Drug: Alprazolam 1mg XR — Alprazolam 1mg XR will be administered for 8 days BID (morning dose only on 8th day)
  Arms: Alprazolam
Drug: Placebo — Placebo, oral tablet/capsule will be administered for 8 days BID (morning dose only on 8th day)
  Arms: Placebo
Drug: CVL-865 low dose — Low dose CVL-865, oral tablets. Will be administered as 2.5mg BID for 2 days followed by 5mg BID for another 2 days during the Titration Phase. 7.5mg BID will be administered during the Maintenance Phase (3 days of BID and morning dose only on 4th day)
  Arms: CVL-865

SUMMARY:
The purpose of this study is to determine anxiolytic effect of multiple doses of CVL-865 using an experimental medicine model of carbon dioxide (CO2) inhalation in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects, ages 18 to 55 years, inclusive, at the time of signing the ICF. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and heart rate measurement, 12-lead ECG, and clinical laboratory tests, as evaluated by the investigator.
* Body mass index of 18.5 to 30.0 kg/m2, inclusive, and a total body weight >50 kg (110 lbs)
* A female subject of childbearing potential who is sexually active with a nonsterilized male partner must agree to use a highly effective method of contraception from signing of informed consent and for 30 days post last dose. A male subject with a pregnant or a nonpregnant partner of childbearing potential must agree to use condom during treatment and until the end of relevant systemic exposure in the male subject for 94 days following the last dose with IMP.
* Capable of giving signed informed consent
* Ability, in the opinion of the investigator, to understand the nature of the trial and comply with protocol requirements, including the prescribed dosage regimens, scheduled visits, laboratory tests, and other trial procedures.
* Defined as sensitive to the anxiogenic effects of double-breath CO2 inhalation

Exclusion Criteria:

* Subjects with a current history of clinically significant cardiovascular pulmonary, gastrointestinal, renal, hepatic, metabolic, hematological, immunological, or neurological disease.
* Subjects with a current or past history of clinically significant respiratory conditions
* Subject with a personal or family history of sickle cell anemia
* Subject with a personal or family history of cerebral aneurysm
* Subjects with a clinically significant current or past personal or family history of any psychiatric disorder as classified by DSM-4 or DSM-5 criteria
* Subjects with epilepsy or a history of seizures except for a single seizure episode
* Subjects with a history of substance or alcohol-use disorder (DSM-5 criteria)
* Subjects who answer "Yes" on the C-SSRS Suicidal Ideation Item 4, 5 and whose most recent episode meeting criteria for this C-SSRS Item 4, 5 occurred within the last 6 months
* Subjects who, in the opinion of the investigator, present a serious risk of suicide
* Subjects with human immunodeficiency virus seropositive status or acquired immunodeficiency syndrome, chronic hepatitis B or C (defined as positive serology and aspartate aminotransferase or alanine aminotransferase elevated to >2 × ULN)
* Subject with a positive drug screen for illicit drugs
* Subjects with a 12-lead ECG demonstrating either of the following:

  * QT interval corrected for heart rate using Fridericia's formula >450 msec (average of 3 ECGs obtained at the Screening Visit)
  * QRS interval >120 msec at the Screening Visit
* Subjects with any of the following abnormalities in clinical laboratory tests at the Screening Visit, as assessed by the local laboratory and confirmed by a single repeat measurement, if deemed necessary:

  * AST or ALT ≥2 × ULN
  * Total bilirubin ≥1.5 × ULN. Subjects with a history of Gilbert's syndrome may be eligible provided the direct bilirubin is <ULN
  * Females: Hemoglobin <11 g/dL; Males: hemoglobin <12 g/dL
  * White blood cell count <3.0 × 109/L
  * Neutrophil count <2.0 × 109/L
  * Platelet count <150 × 109/L
* Subjects with other abnormal laboratory test results, vital sign results, or ECG findings unless, based on the investigator's judgment, the findings are not medically significant
* Systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg at Screening or Day -1
* Subjects taking prohibited medication or who would be likely to require prohibited concomitant therapy
* Subject has a current or past history of BZD abuse and/or dependence
* Female subjects who are breastfeeding and/or who have a positive pregnancy test result prior to receiving IMP
* Subjects who currently use or have used tobacco or nicotine-containing products within 30 days prior to signing the ICF. Subjects who test positive for urine cotinine
* Subjects who has a history of consuming foods or beverages containing >8 units of methylxanthines per day and refuses to abstain from consumption of methylxanthine containing food and beverages while in the clinic.
* Subjects with any condition possibly affecting drug absorption
* Subjects with difficulty swallowing
* Subjects who are known to be allergic or hypersensitive to the IMP or any of its components
* Subjects with a known sensitivity or contraindication to alprazolam
* Subjects who have participated in any clinical trial within 90 days prior to signing the ICF.
* Subjects who have demonstrated a non-response to 35% CO2 double inhalation challenge in a previous trial.
* Any subject who, in the opinion of the sponsor, investigator, or medical monitor, should not participate in the trial
* Subjects with a positive SARS-CoV-2 quantitative PCR test result at Day -1, Period 1 are excluded. Results from subjects reporting a positive SARS-CoV-2 quantitative PCR test result prior to Day -1, Period need to be discussed with the sponsor/medical monitor prior to enrolment of the subject into the trial

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2021-11-14 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
PSL-IV score | up to Day 8
  Change in Panic Symptom List -IV (PSL-IV), a questionnaire including 13 symptoms, each with intensity rating from 0 (not at all) to 4 (very intense), from pre-CO2 to Post CO2 challenge value

SECONDARY OUTCOMES:
VAS Fear score | up to Day 8
  Change in Visual Analog Scale (VAS) value for fear, consisting of a horizontal line 100 mm in length with 0 corresponding to "no fear" and 100 corresponding to "the most fear possible", from pre-CO2 to Post CO2 challenge
CO2 challenge | Screening, Day 1, Day 8
  Change from pre-CO2 to post-CO2 challenge values in Finapres NanoCore Physiological Measurements
Treatment-emergent AEs | From screening to Follow-up Visit
  Treatment-emergent AEs
Suicidality assessed using Columbia - Suicide Severity Rating Scale (C-SSRS) | Screening, Day -1, Day 8
  Suicidality assessed using Columbia - Suicide Severity Rating Scale (C-SSRS) with no/yes (0/1) to each interview question on the occurrence of suicide events or ideation.
CVL-865 (and alprazolam, if appropriate) concentrations | Day 8
Change From Baseline in NeuroCart test battery Score | Screening, Day 1, Day 8
  Psychodynamic effects of CVL-865 will be assessed by means of the NeuroCart test battery (including saccadic eye movements, adaptive tracking, body sway, Quantitative EEG)
Change from Baseline in Bond & Lader Visual Analogue Scale (VAS) | Day 1, Day 8
  Visual Analogue Scale (VAS) is made up of 16 pairs of alternative descriptors of mood and attention at either end. The Bond-Lader of a 10 cm line. Participants will rate their feelings at the time of assessment by indicating the point on the line which best represent their mood. Each item is scored by measuring the position relative to the left hand end of the line and levels of anxiety, sedation, and dysphoria are then calculated from the combined scores of selected items. The score ranges from 0 to 100, with a high score reflecting a high level of anxiety, sedation or dysphoria.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Etienne Jacobs, PhD, MD, Principal Investigator — Centre for Human Drug Research
Locations (1):
- Centre for Human Drug Research, Leiden, Zernikedreef 8, Netherlands

REFERENCES:
- [Background] Atack JR. GABAA receptor alpha2/alpha3 subtype-selective modulators as potential nonsedating anxiolytics. Curr Top Behav Neurosci. 2010;2:331-60. doi: 10.1007/7854_2009_30. PMID 21309116
- [Background] Atack JR, Hallett DJ, Tye S, Wafford KA, Ryan C, Sanabria-Bohorquez SM, Eng WS, Gibson RE, Burns HD, Dawson GR, Carling RW, Street LJ, Pike A, De Lepeleire I, Van Laere K, Bormans G, de Hoon JN, Van Hecken A, McKernan RM, Murphy MG, Hargreaves RJ. Preclinical and clinical pharmacology of TPA023B, a GABAA receptor &alpha;2/&alpha;3 subtype-selective partial agonist. J Psychopharmacol. 2011 Mar;25(3):329-44. doi: 10.1177/0269881109354928. Epub 2010 Feb 15. PMID 20156926
- [Background] Atack JR, Hutson PH, Collinson N, Marshall G, Bentley G, Moyes C, Cook SM, Collins I, Wafford K, McKernan RM, Dawson GR. Anxiogenic properties of an inverse agonist selective for alpha3 subunit-containing GABA A receptors. Br J Pharmacol. 2005 Feb;144(3):357-66. doi: 10.1038/sj.bjp.0706056. PMID 15655523
- [Background] Atack JR, Wafford KA, Tye SJ, Cook SM, Sohal B, Pike A, Sur C, Melillo D, Bristow L, Bromidge F, Ragan I, Kerby J, Street L, Carling R, Castro JL, Whiting P, Dawson GR, McKernan RM. TPA023 [7-(1,1-dimethylethyl)-6-(2-ethyl-2H-1,2,4-triazol-3-ylmethoxy)-3-(2-fluorophenyl)-1,2,4-triazolo[4,3-b]pyridazine], an agonist selective for alpha2- and alpha3-containing GABAA receptors, is a nonsedating anxiolytic in rodents and primates. J Pharmacol Exp Ther. 2006 Jan;316(1):410-22. doi: 10.1124/jpet.105.089920. Epub 2005 Sep 23. PMID 16183706
- [Background] Bailey JE, Dawson GR, Dourish CT, Nutt DJ. Validating the inhalation of 7.5% CO(2) in healthy volunteers as a human experimental medicine: a model of generalized anxiety disorder (GAD). J Psychopharmacol. 2011 Sep;25(9):1192-8. doi: 10.1177/0269881111408455. PMID 21994314
- [Background] Bandelow B, Zohar J, Hollander E, Kasper S, Moller HJ; WFSBP Task Force on Treatment Guidelines for Anxiety, Obsessive-Compulsive and Post-Traumatic Stress Disoders; Zohar J, Hollander E, Kasper S, Moller HJ, Bandelow B, Allgulander C, Ayuso-Gutierrez J, Baldwin DS, Buenvicius R, Cassano G, Fineberg N, Gabriels L, Hindmarch I, Kaiya H, Klein DF, Lader M, Lecrubier Y, Lepine JP, Liebowitz MR, Lopez-Ibor JJ, Marazziti D, Miguel EC, Oh KS, Preter M, Rupprecht R, Sato M, Starcevic V, Stein DJ, van Ameringen M, Vega J. World Federation of Societies of Biological Psychiatry (WFSBP) guidelines for the pharmacological treatment of anxiety, obsessive-compulsive and post-traumatic stress disorders - first revision. World J Biol Psychiatry. 2008;9(4):248-312. doi: 10.1080/15622970802465807. PMID 18949648
- [Background] Bond A, Lader M. The use of analogue scales in rating subjective feelings. Br J Med Psychol. 1974;47:211-8
- [Background] Borland RG, Nicholson AN. Visual motor co-ordination and dynamic visual acuity. Br J Clin Pharmacol. 1984;18 Suppl 1(Suppl 1):69S-72S. doi: 10.1111/j.1365-2125.1984.tb02583.x. PMID 6525331
- [Background] Borland RG, Nicholson AN. Comparison of the residual effects of two benzodiazepines (nitrazepam and flurazepam hydrochloride) and pentobarbitone sodium on human performance. Br J Clin Pharmacol. 1975 Feb;2(1):9-17. doi: 10.1111/j.1365-2125.1975.tb00465.x. PMID 10941
- [Background] Dias R, Sheppard WF, Fradley RL, Garrett EM, Stanley JL, Tye SJ, Goodacre S, Lincoln RJ, Cook SM, Conley R, Hallett D, Humphries AC, Thompson SA, Wafford KA, Street LJ, Castro JL, Whiting PJ, Rosahl TW, Atack JR, McKernan RM, Dawson GR, Reynolds DS. Evidence for a significant role of alpha 3-containing GABAA receptors in mediating the anxiolytic effects of benzodiazepines. J Neurosci. 2005 Nov 16;25(46):10682-8. doi: 10.1523/JNEUROSCI.1166-05.2005. PMID 16291941
- [Background] Hidalgo RB, Davidson JR. Generalized anxiety disorder. An important clinical concern. Med Clin North Am. 2001 May;85(3):691-710. doi: 10.1016/s0025-7125(05)70336-9. PMID 11349480
- [Background] Leibold NK, van den Hove DL, Viechtbauer W, Buchanan GF, Goossens L, Lange I, Knuts I, Lesch KP, Steinbusch HW, Schruers KR. CO2 exposure as translational cross-species experimental model for panic. Transl Psychiatry. 2016 Sep 6;6(9):e885. doi: 10.1038/tp.2016.162. PMID 27598969
- [Background] Low K, Crestani F, Keist R, Benke D, Brunig I, Benson JA, Fritschy JM, Rulicke T, Bluethmann H, Mohler H, Rudolph U. Molecular and neuronal substrate for the selective attenuation of anxiety. Science. 2000 Oct 6;290(5489):131-4. doi: 10.1126/science.290.5489.131. PMID 11021797
- [Background] Morris HV, Dawson GR, Reynolds DS, Atack JR, Stephens DN. Both alpha2 and alpha3 GABAA receptor subtypes mediate the anxiolytic properties of benzodiazepine site ligands in the conditioned emotional response paradigm. Eur J Neurosci. 2006 May;23(9):2495-504. doi: 10.1111/j.1460-9568.2006.04775.x. PMID 16706856
- [Background] Nickolls SA, Gurrell R, van Amerongen G, Kammonen J, Cao L, Brown AR, Stead C, Mead A, Watson C, Hsu C, Owen RM, Pike A, Fish RL, Chen L, Qiu R, Morris ED, Feng G, Whitlock M, Gorman D, van Gerven J, Reynolds DS, Dua P, Butt RP. Pharmacology in translation: the preclinical and early clinical profile of the novel alpha2/3 functionally selective GABAA receptor positive allosteric modulator PF-06372865. Br J Pharmacol. 2018 Feb;175(4):708-725. doi: 10.1111/bph.14119. Epub 2018 Jan 18. PMID 29214652
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] Rudolph U, Crestani F, Benke D, Brunig I, Benson JA, Fritschy JM, Martin JR, Bluethmann H, Mohler H. Benzodiazepine actions mediated by specific gamma-aminobutyric acid(A) receptor subtypes. Nature. 1999 Oct 21;401(6755):796-800. doi: 10.1038/44579. PMID 10548105
- [Background] Salvadore G, Brooks S, Bleys C, Tatikola K, Remmerie B, Jacobs G, et al. The selective Orexin-1 receptor inhibitor JNJ-61393215 decreases subjective anxiety evoked by 35% CO2 inhalation in healthy subjects. Poster presentation at ASCP 2019 Annual Meeting, May 28-31, Scottsdale, Arizona, USA.
- [Background] Simen A, Whitlock M, Qiu R, Miceli J, Zumpano L, Du Metz M, Dua P, Binneman B. An 8-Week, Randomized, Phase 2, Double-Blind, Sequential Parallel-Group Comparison Study of Two Dose Levels of the GABAA Positive Allosteric Modulator PF-06372865 Compared With Placebo as an Adjunctive Treatment in Outpatients With Inadequate Response to Standard of Care for Generalized Anxiety Disorder. J Clin Psychopharmacol. 2019 Jan/Feb;39(1):20-27. doi: 10.1097/JCP.0000000000000997. PMID 30531477
- [Background] Struzik L, Vermani M, Coonerty-Femiano A, Katzman MA. Treatments for generalized anxiety disorder. Expert Rev Neurother. 2004 Mar;4(2):285-94. doi: 10.1586/14737175.4.2.285. PMID 15853570
- [Background] Wittchen HU, Jacobi F. Size and burden of mental disorders in Europe--a critical review and appraisal of 27 studies. Eur Neuropsychopharmacol. 2005 Aug;15(4):357-76. doi: 10.1016/j.euroneuro.2005.04.012. PMID 15961293
- [Background] Wright BM. A simple mechanical ataxia-meter. J Physiol. 1971 Oct;218 Suppl:27P-28P. No abstract available. PMID 5130616
- [Background] van Steveninck AL, Schoemaker HC, Pieters MS, Kroon R, Breimer DD, Cohen AF. A comparison of the sensitivities of adaptive tracking, eye movement analysis and visual analog lines to the effects of incremental doses of temazepam in healthy volunteers. Clin Pharmacol Ther. 1991 Aug;50(2):172-80. doi: 10.1038/clpt.1991.122. PMID 1868679
- [Background] van Steveninck AL, van Berckel BN, Schoemaker RC, Breimer DD, van Gerven JM, Cohen AF. The sensitivity of pharmacodynamic tests for the central nervous system effects of drugs on the effects of sleep deprivation. J Psychopharmacol. 1999;13(1):10-7. doi: 10.1177/026988119901300102. PMID 10221355
- [Background] Yonkers KA, Bruce SE, Dyck IR, Keller MB. Chronicity, relapse, and illness--course of panic disorder, social phobia, and generalized anxiety disorder: findings in men and women from 8 years of follow-up. Depress Anxiety. 2003;17(3):173-9. doi: 10.1002/da.10106. PMID 12768651